CLINICAL TRIAL: NCT01885143
Title: A Case Collection Study for Digital Breast Tomosynthesis (DBT) Using the Senographe Essential
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 101.01-2013-GES-0001
Record Dates: First submitted 2013-06-14; First posted 2013-06-24 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Image Correction
Keywords: Mammography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Artifact Correction: A minimum of 6 subjects will be recruited for the purpose of evaluating artifact correction
  Interventions: Radiation: Digital Breast Tomosynthesis
- Lossy Compression: A minimum of 6 subjects will be recruited for the purpose of evaluating lossy compression
  Interventions: Radiation: Digital Breast Tomosynthesis

INTERVENTIONS:
Radiation: Digital Breast Tomosynthesis
  Other Names: DBT

SUMMARY:
Collect clinical images requested by FDA with GE Breast Tomosynthesis to show they are of acceptable quality as defined in the relevant FDA guidance document before and after artifact correction and in standard screening images. Lossy compression will also be evaluated to demonstrate that images are of acceptable quality when lossy compression is enabled.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent or have a legally authorized representative provide written informed consent
* Female subjects who are 40 years of age or older
* Subject has no history of symptoms and/or physical signs of breast cancer on the side of the targeted breast
* Subject underwent routine Full-Field Digital Mammography (FFDM) which showed one or more abnormalities, including calcifications, and was referred for diagnostic work-up within 4 weeks
* Subject is surgically sterile (must have documentation of bilateral oophorectomy and/or documented hysterectomy), post-menopausal (must have documentation of cessation of menses for greater than one year) or, if of childbearing potential, a documented negative urine pregnancy test within 4 weeks is required.
* Subject breast size is compatible with the dimensions of 24x31 cm of the image detector
* Subject must be in sufficient good health to be able to undergo an examination on mammography equipment as determined by the Investigator

Exclusion Criteria:

* Subject or a legally authorized representative is unable to provide written informed consent
* Clinical assessment and DBT cannot be performed within 4 weeks of screening FFDM examination
* Subject is breast-feeding
* Subject has breast implants or reconstructed breasts
* Subject is undergoing radiotherapy or chemotherapy
* Subject has a history of prior radiotherapy treatment on the side of the targeted breast
* Subject has been previously enrolled in this study
* Subject is participating or has participated in another trial of an investigational product

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the site's population of women recalled for further workup due to abnormalities found on screening Full-field digital Mammography exam.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-08; Primary Completion 2013-10 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
DBT in Senographe Essential is of acceptable quality according to FDA criteria | Phase 1_12 clinical cases read. Maximum time frame for read to result: 2 weeks
  Collect 12 clinical DBT cases with MLO and CC views taken from the Senographe Essential to assess whether the DBT in Senographe Essential is of acceptable quality according to FDA criteria following the clinical evaluation instructions described in Section 9 of the guidance document "Guidance for Industry and FDA Staff: Class II Special Controls Guidance Document: Full-Field Digital Mammography System". Assessment will include review of images with and without artifact correction and with and without lossy compression and findings will be included in PMA submission.

CONTACTS AND LOCATIONS:
Overall Officials: Murray Rebner, MD, Principal Investigator — Beaumont Hospital System
Locations (1):
- Beaumont Hospitals, Royal Oak, Michigan, United States